CLINICAL TRIAL: NCT04122573
Title: Prospective Multicenter Study for Early Evaluation of Acute Chest Pain
Acronym: PEACP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Dongze Li, Lecturer, Clinical Research, West China Hospital
Other Study IDs: WestChinaH1
Record Dates: First submitted 2019-10-06; First posted 2019-10-10 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Chest Pain; Acute Aortic Dissection; Pulmonary Embolism; Acute Myocardial Infarction Type 1; Acute Coronary Syndrome
Keywords: Chest pain; Acute Aortic Dissection; Pulmonary Embolism; Acute Coronary Syndrome; Acute myocardial infarction; Risk stratification; Prognosis; Biomarkers
MeSH Terms: conditions — Chest Pain; Pulmonary Embolism; Acute Coronary Syndrome | interventions — Coronary Angiography; Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Whole blood and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute chest pain: The population in this study are characterized by acute chest pain as the first symptom for consultation within 24 hours.
  Interventions: Diagnostic Test: Coronary angiography; Diagnostic Test: CT angiography of aorta; Diagnostic Test: CT angiography of pulmonary arteries.; Diagnostic Test: Electrocardiogram; Diagnostic Test: Cardiac Troponin

INTERVENTIONS:
Diagnostic Test: Coronary angiography — Acute chest pain patients, suspected acute coronary syndrome, are diagnosed by coronary angiography.
Diagnostic Test: CT angiography of aorta — Acute chest pain patients, suspected acute aortic dissection, are diagnosed by gold standard of CTA.
  Other Names: CTA
Diagnostic Test: CT angiography of pulmonary arteries. — Acute chest pain patients, suspected acute pulmonary embolism, are diagnosed by gold standard of CTA.
  Other Names: CTA
Diagnostic Test: Electrocardiogram — All patients with acute chest pain will subject to ECG examination within 10 minutes of admission, which can quickly screen ST-segment elevation myocardial infarction.
  Other Names: ECG
Diagnostic Test: Cardiac Troponin — Dynamic changes of cardiac troponin I and/or T will be used in the diagnosis of acute myocardial infarction
  Other Names: Biomarkers of myocardial injury

SUMMARY:
In this study, clinical database and blood sample bank of acute chest pain (ACP) will be established at chest pain center of multi-center hospital. To explore new biomarkers and screen clinical indicators with effective risk stratification and prognostic evaluation for ACP through proteomics technology and statistics methods. Risk stratification and short-term and long-term prognostic evaluation models for high-risk ACP will be established using large data analysis.

DETAILED DESCRIPTION:
In this study, acute chest pain (ACP) patients will be selected from chest pain center of nine large tertiary hospitals in China from November 1, 2019 to October 31, 2021. All the selected patients will sign the informed consent.

Patients' characteristics, the first vital signs at the time of consultation, the first arterial blood gas, complete blood count, coagulation markers, blood biochemical results and myocardial injury markers, imaging examinations and electrocardiogram will be collected within 30 minutes at admission. Meanwhile, whole blood and plasma samples will be collected and stored in - 80 ℃ refrigerator. After diagnosis according to the gold standard examination or related guidelines, patients will be admitted to different department for standard treatment. Medication, surgical procedures and complications will be recorded carefully. Plasma and whole blood will be used to detect proteomics and/or genomics biomarkers associated with early evaluation of ACP.

Screening early evaluation indicators using novel protein biomarkers and easy-to-obtain clinical indicators, and establishing evaluation models for high-risk ACP by data analysis methods. Area under the receiver operating characteristic curves (AUROC), net reclassification improvement (NRI), integrated discrimination improvement (IDI) and decision curve analysis (DCA) will be used to evaluate the prediction ability of the model.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18-90 years old;
* The time from onset of symptoms to emergency room is less than 24 hours.

Exclusion Criteria:

* Patients complicate with end-stage neoplastic diseases;
* Pregnant women;
* Patients re-visit during the selection period;
* Patients refuse to participate in this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population in this study is characterized by acute chest pain as the first symptom for consultation. These are mainly Han and Tibetan patients from southwest China. The study population included first-visit and referral patients.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Rate of participants with all-cause death | One year
  Patients die of all causes during hospitalization or follow-up
Rate of participants with cardiovascular death | One year
  Patients die of cardiac and cerebrovascular diseases during hospitalization or follow-up
Rate of participants with major adverse cardiac events (MACEs) | One year
  MACEs include cardiac death, stroke, and recurrent myocardial infarction.
Rate of participants with acute myocardial infarction | Twenty-four hours
  Chest pain patients are diagnosed as acute myocardial infarction based on fourth edition of guidelines for myocardial infarction
Rate of participants with acute pulmonary embolism | Twenty-four hours
  Chest pain patients are diagnosed as acute pulmonary embolism based on CT of pulmonary angiography.
Rate of participants with acute aortic dissection | Twenty-four hours
  Chest pain patients are diagnosed as acute aortic dissection based on CT of aortic angiography.
Rate of participants with acute coronary syndrome | Twenty-four hours
  Chest pain patients are diagnosed as acute coronary syndrome based on European Society of Cardiology (ESC) guidelines.

SECONDARY OUTCOMES:
Rate of participants with ischemia or necrosis of lower limbs | Two weeks
  Patients complicate with ischemia or necrosis of lower limbs during hospitalization
Rate of participants with acute heart failure | Two weeks
  Patients complicate with acute heart failure during hospitalization
Rate of participants with revascularization | Two weeks
  Patients receive revascularization for recurrent angina or myocardial infarction during hospitalization
Rate of participants with consciousness disorder | Two weeks
  Patients complicate with consciousness disorder during hospitalization
Rate of participants with cardiogenic shock | Two weeks
  Patients complicate with cardiogenic shock during hospitalization
Rate of participants with acute kidney injury | Two weeks
  Patients complicate with acute kidney injury during hospitalization
Rate of participants with malignant arrhythmia | Two weeks
  Patients complicate with malignant arrhythmia during hospitalization
Rate of participants with pericardial tamponade | Two weeks
  Patients complicate with pericardial tamponade during hospitalization
Rate of participants with bleeding | One year
  Patients complicate with bleeding
Rate of participants with multiple organ dysfunction syndrome | Two weeks
  Patients complicate with multiple organ dysfunction syndrome during hospitalization
Rate of participants with respiratory failure | Two weeks
  Patients complicate with respiratory failure during hospitalization
Rate of participants with cardiac arrest | Two weeks
  The sudden termination of cardiac ejection function, the disappearance of great artery pulsation and heart sound, and severe ischemia and hypoxia of important organs (such as brain) lead to the termination of life.

OTHER OUTCOMES:
Length of stay | Two weeks
  Time between patient's visit and discharge
Rate of re-admitted participants | Six months
  Re-admission after discharge within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dongze Li, MBBS, Principal Investigator — Emergency Department, West China Hospital, Sichuan University
Locations (9):
- China (9):
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Chengdu Shangjin Nanfu Hospital, Chengdu, Sichuan
  - Sichuan Integrative Medicine Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - People's Hospital of Xindu District, Chengdu, Sichuan
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Panzhihua Central Hospital, Panzhihua, Sichuan
  - Zigong Fourth People's Hospital, Zigong, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
This study will share individual participant data (IPD) including patient characteristics, vital signs, laboratory examinations, imaging examinations, diagnosis, adverse events in hospital and long-term prognosis.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Six months after completion of the test
Access Criteria: IPD will be public accessable via Electronic Data Capture. (ResMan: http://www.medresman.org.)
URL: http://www.medresman.org

REFERENCES:
- [Derived] Li F, Li D, Yu J, Jia Y, Wen J, Li W, Tong Y, Wu J, Wan Z, Cao Y, Zhang Q, Zeng R. Association Between Plasma Ceramides and One-Year Mortality in Patients with Acute Coronary Syndrome: Insight from the PEACP Study. Clin Interv Aging. 2023 Apr 6;18:571-584. doi: 10.2147/CIA.S402253. eCollection 2023. PMID 37050937